CLINICAL TRIAL: NCT03561922
Title: Impact on Daily Life of Patients Using the Subretinal Implant RETINA IMPLANT Alpha AMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer of the investigational device has ceased all business activities
Sponsor: Retina Implant AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RI-FI-2017
Record Dates: First submitted 2018-05-17; First posted 2018-06-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Retinal Degeneration; Inherited Retinal Dystrophy Primarily Involving Sensory Retina
Keywords: Retinal Degeneration; Artificial Vision; Retinal Prosthesis; Subretinal Implant; Inherited Retinal Dystrophy; Vision Restoration; Bionic Eye; Bionic Vision; Retinitis Pigmentosa; Artificial Retina; Retina Implant; Cone-Rod Dystrophy; Choroideremia; Retinopathia Pigmentosa
MeSH Terms: conditions — Retinal Degeneration; Retinitis Pigmentosa; Cone-Rod Dystrophies; Choroideremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RETINA IMPLANT Alpha AMS (Experimental): All participants receive the subretinal device RETINA IMPLANT Alpha AMS
  Interventions: Device: RETINA IMPLANT Alpha AMS

INTERVENTIONS:
Device: RETINA IMPLANT Alpha AMS — Implantation of the subretinal RETINA IMPLANT Alpha AMS

SUMMARY:
This study aims to assess the impact of the subretinal implant RETINA IMPLANT Alpha AMS on the patient's daily life, using validated activities of daily living and questionnaires.

DETAILED DESCRIPTION:
This study aims to assess the impact of the subretinal implant RETINA IMPLANT Alpha AMS on the patient's daily life. In addition, the study will provide additional information about the safety and efficacy of the CE-certified RETINA IMPLANT Alpha AMS. In several studies it has been shown that patients who received this subretinal implant regain visual function to a certain extent and that its use is safe. So far, all assessments of patients with the RETINA IMPLANT Alpha AMS have been done in a controlled environment within the scope of interventional studies where the benefit in daily life has been assessed anecdotally only. Currently, there is no standard method available for an objective assessment of the impact of such devices in daily life of these patients. Hence, the aim of this study is to further assess the impact in daily life with a combination of already validated and newly developed assessments and questionnaires.

This study adheres to the tenets of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 78
2. Willing and able to give written informed consent
3. Hereditary retinal degeneration of the outer retinal layer i.e. photoreceptors (rods & cones)
4. Pseudophakia or aphakia in the eye to be implanted
5. Retinal vessels with remaining perfusion, despite pathological condition
6. Layering of inner retina in the central region present, as shown by Optical Coherence Tomography (OCT)
7. Thickness of the retina sufficient for subretinal surgery as shown by OCT
8. Inner retina still functional (proven e.g. by light perception or electrically evoked phosphenes (EEP))
9. Blindness in both eyes, (no light perception or light perception only)
10. Visual acuity sufficient for reading normal print in earlier life, optically corrected
11. Period of appropriate visual functions at least 12 years / lifetime
12. Willing and able to perform study assessments and training during the full time period of 12 months
13. Motivation to get the best possible results through training and realistic expectations about these as assessed in screening interview

Exclusion Criteria:

1. OCT shows significant retina edema and/or scar tissue within target region for implant
2. Heavy clumped pigmentation at posterior pole or on the planned route of the implantation
3. atrophy of optic nerve or ganglion cells degeneration
4. Any other ophthalmologic disease with relevant effect upon visual function (e.g. glaucoma, optic neuropathies, trauma, diabetic retinopathy, retinal detachment)
5. Deep amblyopia reported earlier in life on eye to be implanted
6. Systemic conditions that might imply considerable risks with regard to the surgical interventions and anesthesia (e.g. cardiovascular/pulmonary diseases, severe metabolic diseases)
7. Acute and severe neurological and/or psychiatric diseases
8. Hyperthyroidism or hypersensitivity to iodine
9. Hypersensitivity to fluorescent dye
10. Women who are pregnant or nursing, or women of childbearing potential who are not willing to use a medically acceptable means of birth control for the duration of the study or women unwilling to perform a pregnancy test before entering the study
11. Participation in another interventional clinical study within the past 30 days

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Change in functional vision | baseline vs. 12 months after implantation
  Instrumental Activities of Daily Living assessed at baseline (prior to implantation) versus one year after implantation

SECONDARY OUTCOMES:
Vision Related Quality of Life - Questionnaire | at baseline and 1, 2.5, 4, 6, 9 and 12 months after implantation (and for longterm review after 18 and 24 months)
  A validated patient reported outcome questionnaire, IVI-VLV, assessed at baseline versus one year after implantation
Visual Function - Questionnaire | at baseline and 1, 2.5, 4, 6, 9 and 12 months after implantation (and for longterm review after 18 and 24 months)
  A validated patient reported outcome questionnaire, ULV-VFQ, assessed at baseline versus one year after implantation
Adverse Events | 2 years
  Number, nature and severity of device-related and implantation-related adverse events
Measure of implant-mediated visual function | 2 years
  Computer test assessed with implant on versus off

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Leveziel, Prof, Study Chair — Centre Hospitalier Universitaire (CHU) de Poitiers, France; Pierre-André Duval, Dr, Principal Investigator — Clinique Saint Jean, Montpellier, France
Locations (2):
- France (2):
  - Clinique Saint Jean, Montpellier, Hérault
  - Centre Hospitalier Universitaire La Milétrie de Poitiers, Poitiers, Vienne

IPD SHARING:
Plan to Share IPD: Undecided
If data are shared, this will only be done in a pseudonymized manner.

REFERENCES:
- [Background] Stingl K, Schippert R, Bartz-Schmidt KU, Besch D, Cottriall CL, Edwards TL, Gekeler F, Greppmaier U, Kiel K, Koitschev A, Kuhlewein L, MacLaren RE, Ramsden JD, Roider J, Rothermel A, Sachs H, Schroder GS, Tode J, Troelenberg N, Zrenner E. Interim Results of a Multicenter Trial with the New Electronic Subretinal Implant Alpha AMS in 15 Patients Blind from Inherited Retinal Degenerations. Front Neurosci. 2017 Aug 23;11:445. doi: 10.3389/fnins.2017.00445. eCollection 2017. PMID 28878616
- [Background] Edwards TL, Cottriall CL, Xue K, Simunovic MP, Ramsden JD, Zrenner E, MacLaren RE. Assessment of the Electronic Retinal Implant Alpha AMS in Restoring Vision to Blind Patients with End-Stage Retinitis Pigmentosa. Ophthalmology. 2018 Mar;125(3):432-443. doi: 10.1016/j.ophtha.2017.09.019. Epub 2017 Oct 27. PMID 29110946
- See also: Retina Implant AG Sponsor homepage — http://www.retina-implant.de